CLINICAL TRIAL: NCT06988319
Title: Psilocybin for Chronic Pelvic Pain (CPP) in Women: A Pilot Feasibility Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland Psychotherapy Clinic, Research, and Training Center (Other)
Responsible Party: Principal Investigator, Lynne Shinto, ND, MPH, Professor of Neurology, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28634; Circle of Giving Foundation (Other: Oregon Health & Science University)
Record Dates: First submitted 2025-05-02; First posted 2025-05-23 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pelvic Pain
Keywords: psilocybin; women; chronic pelvic pain; psilocybin assisted therapy
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Feasibility and Acceptability study to assess safety of a single dose of pharmaceutical grade psilocybin at 25 mg combined with psychotherapy in women with chronic pelvic pain
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single dose psilocybin (25 mg) (Experimental): Single dose of pharmaceutical grade psilocybin (25 mg) with psychotherapy
  Interventions: Drug: Psilocybin (Usona Institute)

INTERVENTIONS:
Drug: Psilocybin (Usona Institute) — Single dose of pharmaceutical grade psilocybin (25 mg) combined with psychotherapy sessions

SUMMARY:
The primary aim is to determine the feasibility of enrolling and 15 women with chronic pelvic pain (CPP) that have failed one conventional for CPP to obtain preliminary safety data on a single administration of a moderate dose of pharmaceutical grade psilocybin (25 mg) in combination with psychotherapy sessions (two pre-dose preparatory and three post-dose integration sessions).

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) presents a significant challenge in healthcare, affecting approximately 15% of women in the United States and incurring annual healthcare costs upwards of $5.8 billion. This condition extends beyond persistent physical discomfort, profoundly impacting mental health and overall quality of life. Central to many chronic pain syndromes, CPP can lead to a heightened state of pain sensitivity known as central sensitization. This condition arises from neuroplastic changes within the central nervous system, leading to structural, functional, and chemical alterations in the brain that enhance neural reactivity, even in the absence of actual physical injuries. Central sensitization is characterized by widespread, multisite hyperalgesia and allodynia. These changes often co-occur with fatigue, mood and cognitive disturbances, sleep disruptions, and multisensory hypersensitivity, complicating the clinical picture and exacerbating the condition's impact on daily functioning.

The use of psilocybin in chronic pain is a paradigm shift from conventional pain therapy where the goal is pain alleviation, to changing a person's relationship with pain, offering a re-alignment or 'reset' of one's view of their pain, this is an innovative approach. To date, there are no psilocybin studies evaluating CPP.

This is a pilot feasibility and safety study to evaluate a single administration of psilocybin (25 mg) in women with CPP who have failed at least one conventional CPP therapy. The study will enroll 15 women, the primary aim is to assess feasibility that will be met when at least 80% of participants complete the study and attend 80% of 11 study visits (9/11 visits). Safety will be assessed by adverse event reports, safety labs, and vitals assessments.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth, age 18-45 years (pre-menopause)
* CPP for at least 6 months or longer with central sensitization, diagnosed by a provider who specializes in CPP (e.g. MD, DO, NP)
* CPP with central sensitization includes endometriosis, adenomyosis, uterine fibroids, pelvic congestion, other pelvic inflammatory diseases, irritable bowel syndrome, inflammatory bladder disorders, myalgias, or any combination of the aforementioned1,3
* Failing at least 1 treatment for CPP. Failed conventional interventions include pharmacotherapy, non-pharmacotherapy (bladder installations, neuromodulation, trigger point injections, anesthetic blocks, surgery), physical therapy, and/or psychotherapy (e.g. Cognitive Behavioral Therapy)
* Participants will be generally healthy with no exclusionary physical or mental health conditions.

Exclusion Criteria:

* Pelvic pain that is not defined as chronic (e.g. acute pelvic or vaginal infections such as sexually transmitted infections, urinary tract infections, pregnancy)
* Have a history of or a current primary psychotic disorder or bipolar disorder type 1
* Current use of lithium.
* Ketamine-assisted therapy within 12 weeks of the baseline visit (V3) or hallucinogen use within 6 months of study enrollment (e.g. psilocybin at a dose of 10 mg or 1 gram mushroom or greater, LSD, MDMA, DMT)
* Cannabis use (THC, CBD). If willing to taper before the baseline visit (V3) the participant can be included.
* A positive urine drug test for illicit substance use
* a score of 5 or greater on the Alcohol Use Disorder Identification Test- Consumption (AUDIT-C) indicating heavy alcohol use
* Suicidal ideation or serious suicide risk as determined by C-SSRS, if baseline score is 4 or greater.
* Uncontrolled hypertension, cardiovascular disease, chronic neurologic disorders (e.g. Parkinson's disease, dementia, multiple sclerosis, epilepsy)
* Have any current problem which, in the opinion of the investigator or study physician, might interfere with participation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Chronic pelvic pain in women that include some gender specific conditions (e.g. endometriosis)
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment and Retention Feasibility | baseline to 1-month post psilocybin dose
  Proportion of eligible participants who complete the study from baseline to 1 month post psilocybin dose
Acceptability | End-of-Study Visit at 1-month post psilocybin dose
  Acceptability will use qualitative data collection to provide information on the benefits and challenges of the intervention using a semi-structured interview.
Number of participants with treatment related adverse events | From enrollment to 1-month post treatment
  Adverse events will be collected using a 12- item adverse events checklist covering all major organ systems will be included to probe for adverse events. The nature of each AE, its severity (mild, moderate, or severe), its likely relationship to study treatment (definite, probable, possible, not related, or unknown), its duration and any necessary treatment modifications or adjustments will be recorded. In addition to recording of AEs,, and labs to assess basic metabolic function (including liver function tests), a complete blood count

SECONDARY OUTCOMES:
Patient-Reported Outcome Measurement Information System (PROMIS) Pain interference Inventory | From enrollment to 1-month post treatment
  Provides a rating on pain's impact on physical, emotional, and social functioning, enjoyment, and quality of life.
Central Sensitization Questionnaire | From enrollment to 1-month post treatment
  Provides a rating to assess symptoms associated with central sensitization (CS) and related conditions. The inventory is divided in two parts: Part A consists of 25 symptoms rated on a Likert scale from 0 (never) to 3 (often), with a total score ranging from 0 to 100, where scores 40 and higher are considered clinically relevant and indicative of a higher degree of CS. Part B screens for prior diagnoses of conditions related to CS, including seven chronic overlapping pain conditions (COPCs) such as irritable bowel syndrome, fibromyalgia, and migraine, as well as three CS-related disorders like anxiety, depression, and neck injury.
Revised Mystical Experience Questionnaire (MEQ 30) | 24-48 hours post psilocybin dose
  Provides a rating to assess phenomenology and intensity of mystical experiences, often in the context of altered states of consciousness, such as those induced by psychedelics.
Challenging Experience Questionnaire | 24-48 hours post psilocybin dose
  Provides a rating to assess difficult or challenging psychological experiences, often in the context of altered states induced by psychedelics. It evaluates seven domains of challenging experiences: fear, grief, physical distress, insanity, isolation, death, and paranoia.
Modified Differential Emotions Scale (mDES) Questionnaire | From enrollment to 1-month post treatment
  Provides a rating to assess positive and negative emotion.
Reactions to Touch Questionnaire | 24-48 hours post psilocybin dose
  Provides a rating to assess a participant reactions to any physical touch between therapist and participant that occurs during the psychedelic sessions.
PTSD Checklist for DSM-5 Questionnaire | From enrollment to 1-month post treatment
  Provides a rating to assess the presence and severity of post-traumatic stress disorder (PTSD) symptoms based on DSM-5 criteria. It consists of 20 items corresponding to the four symptom clusters: re-experiencing, avoidance, negative alterations in cognition and mood, and hyper-arousal. Total score range of 0 to 80, with higher scores indicating greater symptom severity.
Female Sexual Function Questionnaire | From enrollment to 1-month post treatment
  Provides a rating to assess female sexual health: desire, arousal, lubrication, orgasm, satisfaction, and pain, with each domain scored on a scale contributing to a total score indicated of a woman's sexual function.
Expectancy Visual Analogue Scale | Baseline visit
  A simple expectancy visual analogue scale to provide a rating of treatment expectancy that will be used to assess the mediating effects of expectancy on treatment outcomes. How much do you think this treatment will reduce your pelvic pain? none to minimal reduction (0-4 mm), mild reduction (5-44 mm), moderate reduction (45-74 mm), substantial to complete reduction (75-100 mm).
Beck Depression Inventory II | From enrollment to 1-month post treatment
  Provides a rating of depression severity. The score range is 0-63, a higher score reflects more severe depression.
Beck Anxiety Inventory | From enrollment to 1-month post treatment
  Provides a rating of anxiety severity. The score range is 0-63, a higher score reflects more severe anxiety
Self-Compassion Scale - Short Form | From enrollment to 1-month post treatment
  Provides a rating of self-compassion, or responding to one's own failure, suffering or inadequacies with kindness and compassion and recognizing one's own flaws and suffering as part of common human experience
Snaith-Hamilton Pleasure Scale | From enrollment to 1-month post treatment
  Provides a rating of hedonic pleasure capacity in social interactions (sample item: "I would enjoy being with my family or close friends"). Each question is anchored to a time frame of the "past few days" and rated on a 1 (Strongly disagree) - 4 (Strongly agree) scale.
CompACT-15 | From enrollment to 1-month post treatment
  Provides a rating of psychological flexibility: openness to experience (5 items), behavioral awareness (5 items), and valued action (5 items).

OTHER OUTCOMES:
Columbia-Suicide Severity Rating Scale | From enrollment to 1-month post treatment
  A clinician or self-administered tool designed to assess suicidal ideation and behavior. It evaluates the severity and intensity of suicidal thoughts, including wish to die, active suicidal ideation with or without a plan, and preparatory acts. It also captures suicidal behavior such as attempts, interrupted or aborted attempts, and non-suicidal self-injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No